CLINICAL TRIAL: NCT02929121
Title: A Multi-center, Double-blind, Randomized, 24-month Study, to Compare the Efficacy of Doxycycline Once Daily for 6 Weeks Versus Placebo in Improving Filarial Lymphedema Independent of Active Filarial Infection
Brief Title: A 24 Month Study to Compare Efficacy of Doxycycline vs Placebo for Improving Filarial Lymphedema in India
Acronym: LeDoxy-India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Task Force for Global Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Ottesen, Director of the Neglected Tropical Diseases Support Center, The Task Force for Global Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LeDoxy2015_India
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Lymphedema; Lymphatic Filariasis; Filariasis
Keywords: Lymphedema; Lymphatic Filariasis; Filariasis; Doxycycline
MeSH Terms: conditions — Lymphedema; Elephantiasis, Filarial; Filariasis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline (Active Comparator): The Doxycycline treated group will enroll 125 participants. 100 patients with Grades 1-3 lymphedema per study site (based on end point and duration) and up to 25 patients with grade 4-6 lymphedema/per study site. Each patient will receive Doxycycline hyclate 200 mg per day x 6 weeks for patients >50 kg or 100 mg per day for patients <50 kg).
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): The Placebo treated group will enroll 125 participants. 100 patients with Grades 1-3 lymphedema per study site (based on end point and duration) and up to 25 patients with grade 4-6 lymphedema/per study site. Each patient will receive matching tablets containing no active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Once daily tablet for 6 weeks: Doxycycline hyclate 200 mg per day x 6 weeks for patients >50 kg or 100 mg per day for patients <50 kg)
  Other Names: Doxycycline hyclate
  Arms: Doxycycline
Drug: Placebo — Once daily tablet for 6 weeks: matching tablets containing no active ingredients
  Arms: Placebo

SUMMARY:
Current lymphedema management protocols are based on the use of simple measures of hygiene (regular washing with soap and water, skin and nail care), use of topical antibiotics or antifungal agents, exercise and footwear. This is considered the "standard of care" in most endemic countries in the absence of any structured treatment programs. Previous controlled clinical trials and extensive field experience have shown the benefit of these measures in reducing the frequency of attacks of acute dermato-lymphangio-adenitis (ADLA) that drive the progression of lymphedema.

In the present study, the progression of lymphedema in a group of patients who receive a six-week course of doxycycline will be compared with that of a group who receives doxycycline "look-alike" placebo tablets. However, both groups will be enrolled into a standardized "regimen of hygiene" described above. Thus, patients enrolled in the "placebo" group also will receive the current standard of care, and the placebo used in the study will help to identify the benefits of doxycycline on a background of simple hygiene measures. The regimens will be explained to all participants who will be trained to use established standardized methods of hygiene and be effectively applying it prior to the initiation of the drug treatment. In addition, patients will be evaluated at 3, 6, 12 and 24 months.. A common, generic SOP with handouts that describes methods and the training schedule will be used so that similar methods are employed across all sites.

DETAILED DESCRIPTION:
This (LEDOXY) trial is designed as a randomized, controlled, observer-, provider- and patient-blinded multicenter superiority trial with two parallel groups and a primary endpoint of change in grade of lymphedema at 24 months. The population will be stratified according to the Grade (Early Grade 1-3; Late Grade 4-6). Randomization will be performed as block randomization within each center in blocks of (N=4-10) for each of the groups (Early and Late).

The effect of a 6-week course doxycycline on lymphedema without active filarial infection has been demonstrated in a single setting in Africa (Ghana). In order to expand the benefits of this observation, similar studies need to be carried out in other endemic settings. Lymphatic filariasis is endemic in many countries of Africa and Asia that are yet to implement morbidity management programmes. In addition, the components of the proposed hygiene package are likely to vary depending on the availability of material and human resources. The conduct of this trial as a multi-center study will not only allow the evaluation of the efficacy of the drug in a variety of settings but also facilitate its rapid adoption by the respective control programmes of endemic countries, if proven to be useful.

The choice of study sites in endemic countries has been made based on the availability of a) adequate numbers of patients with various grades of lymphedema and b) clinical trial teams familiar with lymphedema management procedures and past experience with similar trials.

All screened patients will be enrolled into a programme of hygiene (described below) and will be required to demonstrate ability to use established standardized methods of hygiene and effectively applying it prior to the initiation of the drug treatment. Eligible patients will be randomized to receive either daily doxycycline or placebo. Doxycycline and placebo will be provided by Medopharm (India). Re-labeling and packaging of the drug and the placebo will be done by Piramal Healthcare, Morpeth, UK.

Additionally, after un-blinding and data analysis, the placebo group will be offered doxycycline treatment if the intervention proves to be more effective in ameliorating LE.

Both doxycycline and placebo will be administered under supervision (directly observed treatment) for 6 weeks. The first dose of doxycycline (two 100 mg tablets for those over 50kg body weight and one 100 mg tablets for those between 40 and 50 kg body weight) or placebo will be given after all the investigations have been completed and informed consent has been obtained and the patient has been initiated into the programme of basic hygiene. Patients will be encouraged to eat before swallowing the tablets whole with a glass of water. Vomited doses will be replaced.

Ideally, patients will be required to come every day to the closest community health center to take their drugs under supervision. Subjects living in villages at a distance from any health center will be treated by the community health care provider or the local caregiver living in this village who will be informed and trained in the possible adverse events related to the drug.

Since some study sites may be village based without a health centre, patients may be treated in their village and required to attend daily at a fixed meeting point. The trial clinician and the research team with the help of trained community health workers will normally administer the treatment. Patients should come to the clinic every week with the patient and collect the drugs for one week. The provider will keep a diary where he or she will mark down the time of intake of the drug. A health worker may make surprise checks at the patient's residence by looking at the diary and also by counting the remaining drugs to estimate compliance.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following at randomization:

1. Age ≥ 14 years and <65 years, male or non-pregnant women of childbearing-potential using an approved, effective method of contraception before, during and for at least 2 weeks after the completion of the active intervention with doxycycline or placebo
2. Able to give informed consent to participate in the trial (forms to be attached)
3. Resident in endemic area for five years or more
4. Body weight >40 kg
5. Lymphedema of a limb Grade 1-6 measured on a 7-point scale. (Appendix 1 for explanation of the grading system (Dreyer G et al. 2002).
6. Ability to use established standardized methods of hygiene and effectively applying it prior to the initiation of the drug treatment
7. No evidence of severe or systemic comorbidities except for features of filarial disease
8. Normal laboratory profile (Appendix 3 investigations and the maximum or minimum limits in the case of hematological abnormalities - Site Specific)
9. Consent to storage of blood samples for study

Exclusion Criteria:

Patients are ineligible to participate in the trial, if patients have any of the following:

1. No lymphedema or lymphedema stage 7
2. Age < 14 years or > 65 years
3. Body weight < 40 kg
4. Pregnant or breastfeeding women
5. Women of childbearing potential not using an agreed method of contraception. (A pregnancy test will be conducted as part of the screening process to exclude pregnancy and repeated at 3 and 8 weeks. In addition, women of childbearing potential will be counseled against pregnancy during the treatment period)
6. Clinical or laboratory evidence of hepatic or renal dysfunction or CNS disease
7. Alcohol or drug abuse
8. History of adverse reactions to doxycycline or other tetracyclines
9. Patient has any situation or condition that may interfere with participation in the study as judged by the clinical investigator

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Lymphadema Grade | 24 months
  Change in lymphedema grade at 24 months compared to baseline

SECONDARY OUTCOMES:
Change in number of acute attacks | 24 months
  Change in number of acute attacks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ottesen, MD, Principal Investigator — The Task Force for Global Health
Locations (1):
- Filariasis Research Unit Govt. T. D. Medical College Hospital, Alappuzha, Kerala, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shenoy RK, Kumaraswami V, Suma TK, Rajan K, Radhakuttyamma G. A double-blind, placebo-controlled study of the efficacy of oral penicillin, diethylcarbamazine or local treatment of the affected limb in preventing acute adenolymphangitis in lymphoedema caused by brugian filariasis. Ann Trop Med Parasitol. 1999 Jun;93(4):367-77. doi: 10.1080/00034989958366. PMID 10656038
- [Result] Mand S, Debrah AY, Klarmann U, Batsa L, Marfo-Debrekyei Y, Kwarteng A, Specht S, Belda-Domene A, Fimmers R, Taylor M, Adjei O, Hoerauf A. Doxycycline improves filarial lymphedema independent of active filarial infection: a randomized controlled trial. Clin Infect Dis. 2012 Sep;55(5):621-30. doi: 10.1093/cid/cis486. Epub 2012 May 18. PMID 22610930
- [Result] Dreyer G, Dreyer P, Noroes J. [Recommendations for the treatment of bancroftian filariasis in symptomless and diseased patients]. Rev Soc Bras Med Trop. 2002 Jan-Feb;35(1):43-50. doi: 10.1590/s0037-86822002000100009. Portuguese. PMID 11873261
- [Derived] Horton J, Klarmann-Schulz U, Stephens M, Budge PJ, Coulibaly Y, Debrah A, Debrah LB, Krishnasastry S, Mwingira U, Ngenya A, Wanji S, Weerasooriya M, Yahathugoda C, Kroidl I, Deathe D, Majewski A, Sullivan S, Mackenzie C, Nutman TB, Shott JP, Weil G, Ottesen E, Hoerauf A. The design and development of a multicentric protocol to investigate the impact of adjunctive doxycycline on the management of peripheral lymphoedema caused by lymphatic filariasis and podoconiosis. Parasit Vectors. 2020 Mar 30;13(1):155. doi: 10.1186/s13071-020-04024-2. PMID 32228663
- See also: The Task Force for Global Health — http://www.taskforce.org/